CLINICAL TRIAL: NCT02417155
Title: Increasing Plasma Adrenaline Levels Through Breathing Techniques - an Explorative Study
Acronym: INADRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: INADRI
Record Dates: First submitted 2014-12-02; First posted 2015-04-15 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Autoimmune Diseases
Keywords: Autonomic Nerve System; Epinephrin; Hyperventilation; Hypoventilation
MeSH Terms: conditions — Autoimmune Diseases; Hyperventilation; Hypoventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- HTR (Experimental): The 'Hoftraining' group (HTR): a group of subjects (n=10) that will be trained extensively by mr. Hof and his team in both hyper/hypoventilation and strength ventilation breathing techniques. Total time training is 8 days.
  Interventions: Behavioral: Hyper/hypoventilation; Behavioral: Strength ventilation
- EIN (Active Comparator): The 'extensive instruction' group (EIN): a group of subjects (n=10) that will receive an extensive instruction course supervised by the research team (in absence of Mr. Hof) in both hyper/hypoventilation and strength ventilation breathing techniques.
  Interventions: Behavioral: Hyper/hypoventilation; Behavioral: Strength ventilation
- STR (Active Comparator): The 'short training' group (STR): a group of subjects (n=10) that will receive only a short training of 1 hour (immediately prior to the study) by Mr. Hof and his team in both hyper/hypoventilation and strength ventilation breathing techniques.
  Interventions: Behavioral: Hyper/hypoventilation; Behavioral: Strength ventilation
- SIN (Active Comparator): The 'short instruction' group (SIN): a group of subjects (n=10) that will receive no training, but only an short instruction course of 1 hour (immediately prior to the study) supervised by the research team (in absence of Mr. Hof) in both hyper/hypoventilation and strength ventilation breathing techniques.
  Interventions: Behavioral: Hyper/hypoventilation; Behavioral: Strength ventilation

INTERVENTIONS:
Behavioral: Hyper/hypoventilation — Subjects are asked to hyperventilate for an average of 30 breaths. Subsequently, the subjects exhaled and hold their breath for approximately 2 minutes ("retention phase"). The duration of breath retention will be entirely at the discretion of the subject himself. Breath retention is followed by a deep inhalation breath, that will be held for 10 s. Subsequently a new cycle of hyper/hypoventilation begins.
Behavioral: Strength ventilation — This exercise consists of deep inhalations and exhalations in which every inhalation and exhalation is followed by breath holding for 10 s, during which the subject tightens all his body muscles.

SUMMARY:
Inflammatory cytokines play a pivotal role in rheumatoid arthritis (RA) and innovative non-pharmacological therapies aimed at limiting cytokine production are highly warranted. Adrenaline, a neurotransmitter of the autonomic sympathetic nervous system, attenuates cytokine production. Along these lines, endogenous modulation of sympathetic activity could limit inflammation and therefore represent a treatment modality that would empower RA patients to exert self-control over disease activity. However, both the autonomic nervous system and the inflammatory response are regarded as systems that cannot be voluntarily influenced. Nevertheless, results from two recent studies demonstrate that this is possible through techniques developed by 'iceman' Wim Hof, namely meditation, exposure to cold, and breathing exercises. Hof himself and healthy volunteers trained by him were able to voluntarily activate the sympathetic nervous system, resulting in adrenaline release and subsequent suppression of the inflammatory response during experimental human endotoxemia (a model of systemic inflammation elicited by administration of lipopolysaccharide [LPS] in healthy volunteers). Interestingly, while having been taught all three techniques, during the endotoxemia experiment the trained subjects (like Hof himself) predominantly practiced the breathing exercises consisting of two different techniques. A 'hyper/hypoventilation' technique, characterized by cycles of hyperventilation followed by breath retention and a 'strength ventilation' technique consisting of deep inhalations and exhalations followed by breath holding. These techniques resulted in intermittent hypoxia and cyclic shifts in acid-base balance. Based on these observations and previous studies, the investigators hypothesize that these breathing techniques account for the increased production of adrenaline and thus for the suppressed inflammatory response but it is unclear which of these two techniques is most important.

DETAILED DESCRIPTION:
The main objective of the study is to compare the increase in plasma adrenaline levels during the two different breathing techniques in a group of healthy volunteers trained by Hof. Also, the investigators investigate whether it is necessary to be trained by Hof and if a relatively short instruction instead of the extensive training is sufficient. Additionally, the investigators want to evaluate the influence of the training and breathing techniques on pain thresholds.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤35 yrs
* Male
* Healthy

Exclusion Criteria:

* Experience with the methods of Wim Hof or other breathing techniques
* Use of any medication
* Smoking
* Use of recreational drugs within 21 days prior to the experiment day
* Use of caffeine or alcohol within 1 day prior to the experimental day.
* Surgery or trauma with significant blood loss or blood donation within 3 months prior to the experimental day.
* Participation in another clinical trial within 3 months prior to the experimental day.
* History, signs, or symptoms of cardiovascular disease
* History of atrial or ventricular arrhythmia
* Hypertension (RR systolic >160 or RR diastolic >90)
* Hypotension (RR systolic <100 or RR diastolic <50)
* Conduction abnormalities on the ECG consisting of a 1st degree atrioventricular block or a complex bundle branch block
* History of asthma, or any other pulmonary disease
* C reactive protein (CRP) > 20 mg/L, White blood count (WBC) > 12x109/L, or clinically significant acute illness, including infections, within 4 weeks before the experimental day.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Concentration of plasma adrenaline within arm 1 | 1 day
  Our primary endpoint is the difference between plasma adrenaline levels during the hyper/hypoventilation technique and the strength ventilation technique within the HTR group.

SECONDARY OUTCOMES:
Concentration of plasma adrenaline within arms 2, 3, 4 | 1 day
  Blood will be collected into chilled lithium-heparin tubes and will immediately be placed on ice and centrifuged at 2.000 x g for 10 min at 4 degrees celsius after which plasma will be stored at -80 degrees celsius until analysis. Plasma adrenaline is measured using High Performance Liquid Chromatography (HPLC) with fluorometric detection. The investigators will compare levels during the hyper/hypoventilation technique and plasma adrenaline levels during the strength ventilation technique within the EIN, STR and SIN groups.
concentration of plasma adrenaline between arms 1, 2, 3, 4 | 1 day
  Blood will be collected into chilled lithium-heparin tubes and will immediately be placed on ice and centrifuged at 2.000 x g for 10 min at 4 degrees celsius after which plasma will be stored at -80 degrees celsius until analysis. Plasma adrenaline is measured using HPLCy with fluorometric detection. The investigators will compare differences in plasma adrenaline levels during hyper/hypoventilation or strength ventilation between HTR, EIN, STR and SIN groups.
Plasma interleukine 10 concentration | 1 day
  EDTA (ethylenediaminetetraacetic acid) anticoagulated blood will centrifuged immediately at 2.000 x g for 10 min at 4 degrees calcium after which plasma will be stored at -80 degrees until analysis. Concentration of [cytokine] will be measured using a simultaneous Luminex assay according to the manufacturer's instructions (Milliplex; Millipore). The investigators will compare differences between hyper/hypoventilation and strength ventilation within HTR, EIN, STR and SIN groups as well as differences during hyper/hypoventilation or strength ventilation between HTR, EIN, and SIN groups.
Body temperature | 1 day
  Body temperature will be measured using an infrared tympanic thermometer (FirstTemp Genius 2; Sherwood Medical). The investigators will compare differences between hyper/hypoventilation and strength ventilation within HTR, EIN, STR and SIN groups as well as differences during hyper/hypoventilation or strength ventilation between HTR, EIN, and SIN groups.
Heart rate, blood pressure | 1 day
  Heart rate will be recorded with a three-lead electrocardiogram on a Philips MP50 patient monitor. The investigators will compare differences between hyper/hypoventilation and strength ventilation within HTR, EIN, STR and SIN groups as well as differences during hyper/hypoventilation or strength ventilation between HTR, EIN, and SIN groups.
Blood pressure | 1 day
  Blood pressure will be measured on a Philips MP50 patient monitor through a 20-gauge arterial catheter. The investigators will compare differences between hyper/hypoventilation and strength ventilation within HTR, EIN, STR and SIN groups as well as differences during hyper/hypoventilation or strength ventilation between HTR, EIN, and SIN groups.
Leukocyte counts and differentiation | 1 day
  Analysis of leukocyte counts and differentiation will be performed in EDTA anticoagulated blood using routine analysis methods also used for patient samples (flow cytometric analysis on a Sysmex XE-5000). The investigators will compare differences between hyper/hypoventilation and strength ventilation within HTR, EIN, STR and SIN groups as well as differences during hyper/hypoventilation or strength ventilation between HTR, EIN, and SIN groups.
Cortisol (plasma) | 1 day
  Blood will be collected in serum-separating tubes and allowed to clot at room temperature for a minimum of 30 min. Subsequently, samples are centrifuged at 2,000 × g for 10 min at 4 °C, after which serum is stored at -80 °C until analysis. Cortisol levels will be determined using a routine analysis method also used for patient samples (electrochemiluminescent immunoassay on a Modular Analytics E170 (Roche Diagnostics). The investigators will compare differences between hyper/hypoventilation and strength ventilation within HTR, EIN, STR and SIN groups as well as differences during hyper/hypoventilation or strength ventilation between HTR, EIN, and SIN groups.
Noradrenaline | 1 day
  Blood will be collected into chilled lithium-heparin tubes and will immediately be placed on ice and centrifuged at 2.000 x g for 10 min at 4 degrees celsius after which plasma will be stored at -80 degrees celsius until analysis. Plasma noradrenaline is measured using HPLCy with fluorometric detection. The investigators will compare differences between hyper/hypoventilation and strength ventilation within HTR, EIN, STR and SIN groups as well as differences during hyper/hypoventilation or strength ventilation between HTR, EIN, and SIN groups.
Blood gas parameters | 1 day
  Blood gas parameters are analyzed in lithium heparin anticoagulated arterial blood using CG4+ cartridges and a point-of-care i-STAT blood gas analyzer (Abbott). The investigators will compare differences between hyper/hypoventilation and strength ventilation within HTR, EIN, STR and SIN groups as well as differences during hyper/hypoventilation or strength ventilation between HTR, EIN, and SIN groups.
Pain threshold | 1 day
  Pain thresholds before start training/instruction, during each of the breathing techniques, and at the end of the experimental day, objectified with Quantitive Sensory Testing by a dedicated, trained member of the studyteam.

CONTACTS AND LOCATIONS:
Overall Officials: Matthijs Kox, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Intensive Care Medicine, Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Background] Kox M, van Eijk LT, Zwaag J, van den Wildenberg J, Sweep FC, van der Hoeven JG, Pickkers P. Voluntary activation of the sympathetic nervous system and attenuation of the innate immune response in humans. Proc Natl Acad Sci U S A. 2014 May 20;111(20):7379-84. doi: 10.1073/pnas.1322174111. Epub 2014 May 5. PMID 24799686
- [Background] Kox M, Stoffels M, Smeekens SP, van Alfen N, Gomes M, Eijsvogels TM, Hopman MT, van der Hoeven JG, Netea MG, Pickkers P. The influence of concentration/meditation on autonomic nervous system activity and the innate immune response: a case study. Psychosom Med. 2012 Jun;74(5):489-94. doi: 10.1097/PSY.0b013e3182583c6d. PMID 22685240
- [Derived] Zwaag J, Naaktgeboren R, van Herwaarden AE, Pickkers P, Kox M. The Effects of Cold Exposure Training and a Breathing Exercise on the Inflammatory Response in Humans: A Pilot Study. Psychosom Med. 2022 May 1;84(4):457-467. doi: 10.1097/PSY.0000000000001065. Epub 2022 Feb 23. PMID 35213875